CLINICAL TRIAL: NCT00533949
Title: A Randomized Phase III Comparison of Standard-Dose (60 Gy) Versus High-Dose (74 Gy) Conformal Radiotherapy With Concurrent and Consolidation Carboplatin/Paclitaxel +/- Cetuximab (IND #103444) in Patients With Stage IIIA/IIIB Non-Small Cell Lung Cancer
Brief Title: High-Dose or Standard-Dose Radiation Therapy and Chemotherapy With or Without Cetuximab in Treating Patients With Newly Diagnosed Stage III Non-Small Cell Lung Cancer That Cannot Be Removed by Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Radiation Therapy Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH); North Central Cancer Treatment Group (Network); Cancer and Leukemia Group B (Network); NRG Oncology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: RTOG 0617; CDR0000564240; NCCTG-N0628; CALGB-30609; NCI-2013-01762 (Registry Identifier: CTRP (Clinical Trials Reporting Program))
Record Dates: First submitted 2007-09-20; First posted 2007-09-24 (Estimated); Results first posted 2017-05-05 (Actual); Last update posted 2022-06-21 (Actual); Status verified 2022-05

CONDITIONS: Lung Cancer; Radiation Toxicity
Keywords: radiation toxicity; stage IIIA non-small cell lung cancer; stage IIIB non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Radiation Injuries; Carcinoma, Non-Small-Cell Lung | interventions — Cetuximab; Carboplatin; Paclitaxel; Albumin-Bound Paclitaxel

STUDY DESIGN:
Intervention Model Description: This study was revised 06/18/08 to a 2x2 factorial design to evaluate the addition of cetuximab to the radiation therapy regimens.
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 60 Gy RT (Active Comparator): 60 Gy Radiation therapy with concurrent paclitaxel and carboplatin followed by consolidation paclitaxel and carboplatin
  Interventions: Drug: Carboplatin; Drug: Paclitaxel; Radiation: 60 Gy RT
- 74 Gy RT (Experimental): 74 Gy Radiation therapy with concurrent paclitaxel and carboplatin followed by consolidation paclitaxel and carboplatin
  Interventions: Drug: Carboplatin; Drug: Paclitaxel; Radiation: 74 Gy RT
- 60 Gy RT + Cetuximab (Experimental): 60 Gy Radiation therapy with concurrent cetuximab, paclitaxel, and carboplatin followed by consolidation cetuximab, paclitaxel, and carboplatin
  Interventions: Biological: Cetuximab; Drug: Carboplatin; Drug: Paclitaxel; Radiation: 60 Gy RT
- 74 Gy RT + Cetuximab (Experimental): 74 Gy Radiation therapy with concurrent cetuximab, paclitaxel, and carboplatin followed by consolidation cetuximab, paclitaxel, and carboplatin
  Interventions: Biological: Cetuximab; Drug: Carboplatin; Drug: Paclitaxel; Radiation: 74 Gy RT

INTERVENTIONS:
Biological: Cetuximab — Loading dose: 400 mg/m2, IV, one week prior to start of radiation therapy (RT). Then, beginning day 1 of RT, 250 mg/m2, IV, weekly; for 60 Gy arm for 15 weeks, for 74 Gy arm for 16 weeks.
  Other Names: Erbitux
  Arms: 60 Gy RT + Cetuximab; 74 Gy RT + Cetuximab
Drug: Carboplatin — Concurrent: AUC=2, IV, days 1, 8, 14, 22, 29, and 36 of radiation therapy; for 74 Gy arms, on day 43 as well.
  Consolidation, 3 weeks after completion of RT, AUC=6, IV, days 1 and 22.
  Other Names: Paraplatin
Drug: Paclitaxel — Concurrent: 45 mg/m2, IV, days 1, 8, 14, 22, 29, and 36 of radiation therapy (RT); for 74 Gy arms, on day 43 as well.
  Consolidation, 3 weeks after completion of RT, 200 mg/m2, IV, days 1 and 22.
  Other Names: Taxol; Abraxane
Radiation: 60 Gy RT — Radiation therapy (RT) in once-daily, 2 Gy fractions, given in 30 fractions over the course of 6 weeks.
  Other Names: RT
  Arms: 60 Gy RT; 60 Gy RT + Cetuximab
Radiation: 74 Gy RT — Radiation therapy (RT) in once-daily, 2 Gy fractions, given in 37 fractions over the course of 7.5 weeks.
  Arms: 74 Gy RT; 74 Gy RT + Cetuximab

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to kill tumor cells. Drugs used in chemotherapy, such as paclitaxel, carboplatin work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Monoclonal antibodies, such as cetuximab can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. It is not yet known whether high-dose radiation therapy is more effective than standard-dose radiation therapy when given together with combination chemotherapy with or without cetuximab in treating patients with non-small cell lung cancer.

PURPOSE: This randomized phase III trial is studying high-dose or standard-dose radiation therapy given together with chemotherapy with or without cetuximab to see how well they work in treating patients with newly diagnosed stage III non-small cell lung cancer that cannot be removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To compare the overall survival of patients with newly diagnosed, unresectable stage IIIA or IIIB non-small cell lung cancer treated with high- versus standard-dose conformal radiotherapy with concurrent and consolidation chemotherapy comprising carboplatin and paclitaxel.
* To compare the overall survival of patients treated with versus without cetuximab in the setting of concurrent chemotherapy

Secondary

* To compare progression-free survival and local-regional tumor control in patients treated with these regimens.
* To compare the toxicity of high- versus standard-dose conformal radiotherapy and concurrent chemotherapy with versus without cetuximab in these patients.
* To investigate the prognostic and predictive effects of gross tumor volume on overall survival of patients treated with these regimens.
* To compare the quality of life of patients treated with these regimens.
* To correlate outcomes (i.e., survival, toxicity, or QOL) in these patients with biological parameters.
* To analyze the predictive value of pre-treatment standardized uptake value (SUV) of positron emission tomography (PET) scan in predicting survival, distant metastasis, and local-regional control in patients treated with these regimens.
* To explore biological markers to predict clinical outcome including survival, distant metastasis, local-regional control, and QOL (including toxicity) in patients treated with these regimens.
* To prospectively collect and bank tissue, blood, and urine specimens for future biomarker analyses in predicting clinical outcome in patients treated with these regimens.
* To investigate associations between epidermal growth factor receptor (EGFR) expression and toxicity, response, overall survival, and progression-free survival.

OUTLINE: This is a multicenter study. Patients are stratified according to PET staging (yes vs no), radiotherapy technique (3-dimensional conformal radiotherapy vs intensity-modulated radiotherapy), Zubrod performance status (0 vs 1), and histology (squamous vs non-squamous). Patients are randomized to 1 of 4 treatment arms. (Arms II and IV closed to accrual effective 6/17/11)

Patients may undergo tumor tissue, blood, and urine collection periodically during study for tissue banking or biomarker correlative studies.

Patients may undergo quality-of-life assessment at baseline and periodically during study.

After completion of study therapy, patients are followed periodically for 5 years and then annually thereafter.

ELIGIBILITY:
Inclusion criteria:

1. Pathologically proven (either histologic or cytologic) diagnosis of Stage IIIA or IIIB non-small cell lung cancer (NSCLC); excluding patients with N3 disease based on supraclavicular or contralateral hilar adenopathy, [according to American Joint Committee on Cancer (AJCC) Staging, 6th edition; see appendix III] within 12 weeks of registration; patients who present with N2 or N3 disease and an undetectable NSCLC primary tumor also are eligible.
2. Patients must be considered unresectable or inoperable; Note: Patients who have had a nodal recurrence after surgery for an early-stage NSCLC are eligible if the following criteria are met:

   * Nodal recurrence must be N1 or N2; N3 is not eligible.
   * The initial primary must have been staged as T1-2, N0, M0.
   * The node must be biopsied within 12 weeks of registration.
   * The node must be measurable.
   * The patient must not have received prior chemotherapy or radiation for this lung cancer.
   * Prior curative surgery must have been at least 6 months prior to the nodal recurrence.
   * The exception to a prior invasive malignancy does not apply to the initial lung primary.
3. Stage III A or B disease, including no distant metastases, based upon the following minimum diagnostic workup are acceptable:

   * History/physical examination, including documentation of height, weight, body surface area (BSA), and vital signs within 8 weeks prior to registration;
   * Computed tomographic (CT)/Magnetic Resonance Imaging (MRI) imaging of the lung and upper abdomen through the adrenal glands within 6 weeks prior to registration;
   * An MRI of the brain with contrast (or CT with contrast if MRI is medically contraindicated) within 6 weeks prior to registration; Note: The use of intravenous contrast is required for the MRI or CT. An MRI without contrast is only permitted if the patient has a contrast allergy.
   * Whole-body fluorodeoxyglucose (FDG) - Positron Emission Tomography(PET) or PET/CT or if no PET is available, a bone scan is required within 6 weeks prior to registration; Note: If a PET is done that shows clear adrenals and lungs, then a CT scan of chest only is permitted.
4. If a pleural effusion is present, the following criteria must be met to exclude malignant involvement (incurable T4 disease):

   * When pleural fluid is visible on both the CT scan and on a chest x-ray, a pleuracentesis is required to confirm that the pleural fluid is cytologically negative.
   * Exudative pleural effusions are excluded, regardless of cytology;
   * Effusions that are minimal (i.e. not visible on chest x-ray) that are too small to safely tap are eligible.
5. Patients must have measurable or evaluable disease.
6. Patients with post-obstructive pneumonia are eligible.
7. Patients must be at least 3 weeks from prior thoracotomy (if performed).
8. Zubrod Performance Status 0-1;
9. Age ≥ 18;
10. Pulmonary function tests (PFTs) including forced expiratory volume in one second (FEV1) within 12 weeks prior to registration; for FEV1, the best value obtained pre- or post bronchodilator must be ≥ 1.2 liters/second or ≥ 50% predicted.
11. Complete blood count (CBC)/differential obtained within 2 weeks prior to registration on study, with adequate bone marrow function defined as follows:

    * Absolute neutrophil count (ANC) ≥ 1,800 cells/mm3;
    * Platelets ≥ 100,000 cells/mm3;
    * Hemoglobin ≥ 10.0 g/dl (Note: The use of transfusion or other intervention to achieve Hgb ≥ 10.0 g/dl is acceptable.)
12. Serum creatinine within normal institutional limits or creatinine clearance ≥60 ml/min;
13. Bilirubin must be within or below normal institutional limits;
14. Aspartate aminotransferase (AST) and Alanine aminotransferase (ALT) < 2.5 x the institutional upper limit of normal (IULN);
15. Patient must sign study specific informed consent prior to study entry.

Exclusion Criteria:

1. N3 supraclavicular disease;
2. Greater than minimal, exudative, or cytologically positive pleural effusions;
3. Involved contralateral hilar nodes (i.e. greater than 1.5 cm on short axis or positive on PET scan);
4. ≥ 10% weight loss within the past month;
5. Prior invasive malignancy (except non-melanomatous skin cancer) unless disease free for a minimum of 3 years; non-invasive conditions such as carcinoma in situ of the breast, oral cavity, or cervix are all permissible.
6. Prior systemic chemotherapy for the study cancer; note that prior chemotherapy for a different cancer is allowable.
7. Prior radiotherapy to the region of the study cancer that would result in overlap of radiation therapy fields;
8. Prior therapy that specifically and directly targets the epidermal growth factor receptor (EGFR) pathway;
9. Prior severe infusion reaction to a monoclonal antibody;
10. Severe, active co-morbidity, defined as follows:

    * Significant history of uncontrolled cardiac disease; i.e., uncontrolled hypertension, unstable angina, myocardial infarction within the last 6 months, uncontrolled congestive heart failure, and cardiomyopathy with decreased ejection fraction.
    * Transmural myocardial infarction within the last 6 months;
    * Acute bacterial or fungal infection requiring intravenous antibiotics at the time of registration;
    * Chronic Obstructive Pulmonary Disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy within 30 days before registration;
    * Hepatic insufficiency resulting in clinical jaundice and/or coagulation defects;
    * Acquired Immune Deficiency Syndrome (AIDS) based upon current Centers for Disease Control and Prevention (CDC) definition; note, however, that human immunodeficiency virus (HIV) testing is not required for entry into this protocol. The need to exclude patients with AIDS from this protocol is necessary because the treatments involved in this protocol may be significantly immunosuppressive. Protocol-specific requirements may also exclude immuno-compromised patients.
11. Pregnancy or women of childbearing potential and men who are sexually active and not willing/able to use medically acceptable forms of contraception; this exclusion is necessary because the treatment involved in this study may be significantly teratogenic.
12. Any history of allergic reaction to paclitaxel or other taxanes, or to carboplatin;
13. Uncontrolled neuropathy grade 2 or greater regardless of cause.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 544 (Actual)
Dates: Start 2007-11; Primary Completion 2013-06 (Actual); Study Completion 2022-05-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Bradley, MD, Principal Investigator — Mallinckrodt Institute of Radiology at Washington University Medical Center; Hak Choy, MD, Study Chair — Simmons Cancer Center; Gregory A. Masters, MD, Study Chair — CCOP - Christiana Care Health Services; Steven E. Schild, MD, Study Chair — Mayo Clinic; Alex A. Adjei, MD, PhD, Study Chair — Roswell Park Cancer Institute; Jeffrey A. Bogart, MD, Study Chair — State University of New York - Upstate Medical University; Arthur William Blackstock, MD, Study Chair — Wake Forest University Health Sciences; Mark A. Socinski, MD, Study Chair — UNC Lineberger Comprehensive Cancer Center; George Blumenschein, MD, Study Chair — M.D. Anderson Cancer Center; Ritsuko Komaki, MD, Study Chair — M.D. Anderson Cancer Center; Jeff Sloan, PhD, HSR, Study Chair — Mayo Clinic; Mark Dobelbower, MD PhD, Study Chair — University of Alabama Medical Center; Tien Hoang, MD, Study Chair — University of Wisconsin, Madison; Ken Forster, PhD, Study Chair — H. Lee Moffitt Cancer Center; Benjamin Movsas, MD, Study Chair — Henry Ford Hospital; Joe Y. Chang, MD PhD, Study Chair — M.D. Anderson Cancer Center; Joseph O. Deasy, PhD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (213):
- United States (207):
  - UAB Comprehensive Cancer Center, Birmingham, Alabama
  - Mayo Clinic Scottsdale, Scottsdale, Arizona
  - Arizona Oncology - Tucson, Tucson, Arizona
  - Mercy Cancer Center at Mercy San Juan Medical Center, Carmichael, California
  - Enloe Cancer Center at Enloe Medical Center, Chico, California
  - Cancer Care Center at John Muir Health - Concord Campus, Concord, California
  - Saint Agnes Cancer Center at Saint Agnes Medical Center, Fresno, California
  - Rebecca and John Moores UCSD Cancer Center, La Jolla, California
  - Memorial Medical Center, Modesto, California
  - St. Joseph Hospital Regional Cancer Center - Orange, Orange, California
  - Feather River Hospital Cancer Center, Paradise, California
  - Radiation Oncology Center - Roseville, Roseville, California
  - Radiological Associates of Sacramento Medical Group, Incorporated, Sacramento, California
  - University of California Davis Cancer Center, Sacramento, California
  - UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - Saint Helena Hospital, St. Helena, California
  - Stanford Cancer Center, Stanford, California
  - Penrose Cancer Center at Penrose Hospital, Colorado Springs, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Poudre Valley Radiation Oncology, Fort Collins, Colorado
  - North Suburban Medical Center, Thornton, Colorado
  - CCOP - Christiana Care Health Services, Newark, Delaware
  - Washington Cancer Institute at Washington Hospital Center, Washington D.C., District of Columbia
  - Broward General Medical Center Cancer Center, Fort Lauderdale, Florida
  - University of Florida Shands Cancer Center, Gainesville, Florida
  - Memorial Cancer Institute at Memorial Regional Hospital, Hollywood, Florida
  - Baptist Cancer Institute - Jacksonville, Jacksonville, Florida
  - Integrated Community Oncology Network at Southside Cancer Center, Jacksonville, Florida
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - Baptist Medical Center South, Jacksonville, Florida
  - Integrated Community Oncology Network, Jacksonville Beach, Florida
  - Ella Milbank Foshay Cancer Center at Jupiter Medical Center, Jupiter, Florida
  - Baptist-South Miami Regional Cancer Program, Miami, Florida
  - CCOP - Mount Sinai Medical Center, Miami Beach, Florida
  - Integrated Community Oncology Network - Orange Park, Orange Park, Florida
  - M.D. Anderson Cancer Center at Orlando, Orlando, Florida
  - Florida Cancer Center - Palatka, Palatka, Florida
  - Sacred Heart Cancer Center at Sacred Heart Hospital, Pensacola, Florida
  - Flagler Cancer Center, Saint Augustine, Florida
  - Georgia Cancer Center for Excellence at Grady Memorial Hospital, Atlanta, Georgia
  - Emory Crawford Long Hospital, Atlanta, Georgia
  - Piedmont Hospital, Atlanta, Georgia
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - Charles B. Eberhart Cancer Center at DeKalb Medical Center, Decatur, Georgia
  - Saint Alphonsus Cancer Care Center at Saint Alphonsus Regional Medical Center, Boise, Idaho
  - Mountain States Tumor Institute at St. Luke's Regional Medical Center, Boise, Idaho
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Creticos Cancer Center at Advocate Illinois Masonic Medical Center, Chicago, Illinois
  - Community Cancer Center, Normal, Illinois
  - Cancer Treatment Center at Pekin Hospital, Pekin, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF St. Francis Medical Center, Peoria, Illinois
  - Radiation Oncology Associates Southwest, Fort Wayne, Indiana
  - Parkview Regional Cancer Center at Parkview Health, Fort Wayne, Indiana
  - Center for Cancer Care at Goshen General Hospital, Goshen, Indiana
  - Central Indiana Cancer Centers - East, Indianapolis, Indiana
  - Community Regional Cancer Care at Community Hospital East, Indianapolis, Indiana
  - Community Regional Cancer Care at Community Hospital North, Indianapolis, Indiana
  - Cancer Center at Ball Memorial Hospital, Muncie, Indiana
  - Mercy Regional Cancer Center at Mercy Medical Center, Cedar Rapids, Iowa
  - John Stoddard Cancer Center at Iowa Methodist Medical Center, Des Moines, Iowa
  - Mercy Cancer Center at Mercy Medical Center - Des Moines, Des Moines, Iowa
  - Mercy Cancer Center at Mercy Medical Center - North Iowa, Mason City, Iowa
  - Siouxland Hematology-Oncology Associates, LLP, Sioux City, Iowa
  - Central Baptist Hospital, Lexington, Kentucky
  - Tulane Cancer Center Office of Clinical Research, Alexandria, Louisiana
  - Mary Bird Perkins Cancer Center - Baton Rouge, Baton Rouge, Louisiana
  - MBCCOP - LSU Health Sciences Center, New Orleans, Louisiana
  - CCOP - Ochsner, New Orleans, Louisiana
  - Greenebaum Cancer Center at University of Maryland Medical Center, Baltimore, Maryland
  - St. Agnes Hospital Cancer Center, Baltimore, Maryland
  - Shore Regional Cancer Center at Memorial Hospital - Easton, Easton, Maryland
  - Peninsula Regional Medical Center, Salisbury, Maryland
  - Baystate Regional Cancer Program at D'Amour Center for Cancer Care, Springfield, Massachusetts
  - Saint Joseph Mercy Cancer Center, Ann Arbor, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Josephine Ford Cancer Center at Henry Ford Hospital, Detroit, Michigan
  - Lacks Cancer Center at Saint Mary's Health Care, Grand Rapids, Michigan
  - Van Elslander Cancer Center at St. John Hospital and Medical Center, Grosse Pointe Woods, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - St. Mary Mercy Hospital, Livonia, Michigan
  - Mercy Regional Cancer Center at Mercy Hospital, Port Huron, Michigan
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Minnesota Oncology Hematology, PA - Maplewood, Maplewood, Minnesota
  - Virginia Piper Cancer Institute at Abbott - Northwestern Hospital, Minneapolis, Minnesota
  - Humphrey Cancer Center at North Memorial Outpatient Center, Robbinsdale, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CentraCare Clinic - River Campus, Saint Cloud, Minnesota
  - Regions Hospital Cancer Care Center, Saint Paul, Minnesota
  - University of Mississippi Cancer Clinic, Jackson, Mississippi
  - Regional Cancer Center at Singing River Hospital, Pascagoula, Mississippi
  - Siteman Cancer Center at Barnes-Jewish St. Peters Hospital - St. Peters, City of Saint Peters, Missouri
  - Siteman Cancer Center at Barnes-Jewish Hospital - Saint Louis, St Louis, Missouri
  - Barnes-Jewish West County Hospital, St Louis, Missouri
  - Billings Clinic - Downtown, Billings, Montana
  - Good Samaritan Cancer Center at Good Samaritan Hospital, Kearney, Nebraska
  - Saint Elizabeth Cancer Institute at Saint Elizabeth Regional Medical Center, Lincoln, Nebraska
  - Methodist Estabrook Cancer Center, Omaha, Nebraska
  - CCOP - Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Renown Institute for Cancer at Renown Regional Medical Center, Reno, Nevada
  - Saint Mary's Regional Medical Center, Reno, Nevada
  - Payson Center for Cancer Care at Concord Hospital, Concord, New Hampshire
  - Center for Cancer Care at Exeter Hospital, Exeter, New Hampshire
  - Elliot Regional Cancer Center at Elliot Hospital, Manchester, New Hampshire
  - Fox Chase Virtua Health Cancer Program at Virtua Memorial Hospital Marlton, Marlton, New Jersey
  - UMDNJ University Hospital, Newark, New Jersey
  - J. Phillip Citta Regional Cancer Center at Community Medical Center, Toms River, New Jersey
  - Cancer Institute of New Jersey at Cooper - Voorhees, Voorhees Township, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - New York Oncology Hematology, PC at Albany Regional Cancer Care, Albany, New York
  - Veterans Affairs Medical Center - Albany, Albany, New York
  - Sands Cancer Center, Canandaigua, New York
  - St. Luke's - Roosevelt Hospital Center - St.Luke's Division, New York, New York
  - Highland Hospital of Rochester, Rochester, New York
  - University Radiation Oncology at Parkridge Hospital, Rochester, New York
  - James P. Wilmot Cancer Center at University of Rochester Medical Center, Rochester, New York
  - SUNY Upstate Medical University Hospital, Syracuse, New York
  - Alamance Cancer Center at Alamance Regional Medical Center, Burlington, North Carolina
  - Lineberger Comprehensive Cancer Center at University of North Carolina - Chapel Hill, Chapel Hill, North Carolina
  - Blumenthal Cancer Center at Carolinas Medical Center, Charlotte, North Carolina
  - Presbyterian Cancer Center at Presbyterian Hospital, Charlotte, North Carolina
  - Kinston Medical Specialists, Kinston, North Carolina
  - FirstHealth Moore Regional Community Hospital Comprehensive Cancer Center, Pinehurst, North Carolina
  - Cancer Centers of North Carolina - Raleigh, Raleigh, North Carolina
  - CCOP - MeritCare Hospital, Fargo, North Dakota
  - Altru Cancer Center at Altru Hospital, Grand Forks, North Dakota
  - Trinity CancerCare Center, Minot, North Dakota
  - McDowell Cancer Center at Akron General Medical Center, Akron, Ohio
  - Summa Center for Cancer Care at Akron City Hospital, Akron, Ohio
  - Barberton Citizens Hospital, Barberton, Ohio
  - Aultman Cancer Center at Aultman Hospital, Canton, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Charles M. Barrett Cancer Center at University Hospital, Cincinnati, Ohio
  - Case Comprehensive Cancer Center, Cleveland, Ohio
  - Cleveland Clinic Cancer Center at Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Riverside Methodist Hospital Cancer Care, Columbus, Ohio
  - Cleveland Clinic Cancer Center, Independence, Ohio
  - Hillcrest Cancer Center at Hillcrest Hospital, Mayfield Heights, Ohio
  - Southwest General Health Center, Middleburg Heights, Ohio
  - UHHS Chagrin Highlands Medical Center, Orange, Ohio
  - St. Charles Mercy Hospital, Oregon, Ohio
  - North Coast Cancer Care, Incorporated, Sandusky, Ohio
  - Flower Hospital Cancer Center, Sylvania, Ohio
  - St. Anne Mercy Hospital, Toledo, Ohio
  - UHHS Westlake Medical Center, Westlake, Ohio
  - Cleveland Clinic - Wooster, Wooster, Ohio
  - Oklahoma University Cancer Institute, Oklahoma City, Oklahoma
  - Natalie Warren Bryant Cancer Center at St. Francis Hospital, Tulsa, Oklahoma
  - Willamette Valley Cancer Center - Eugene, Eugene, Oregon
  - Morgan Cancer Center at Lehigh Valley Hospital - Cedar Crest, Allentown, Pennsylvania
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Geisinger Cancer Institute at Geisinger Health, Danville, Pennsylvania
  - Northeast Radiation Oncology Center, Dunmore, Pennsylvania
  - Dale and Frances Hughes Cancer Center at Pocono Medical Center, East Stroudsburg, Pennsylvania
  - Regional Cancer Center - Erie, Erie, Pennsylvania
  - Penn State Hershey Cancer Institute at Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Cancer Center of Paoli Memorial Hospital, Paoli, Pennsylvania
  - Kimmel Cancer Center at Thomas Jefferson University - Philadelphia, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center - Philadelphia, Philadelphia, Pennsylvania
  - Frankford Hospital Cancer Center - Torresdale Campus, Philadelphia, Pennsylvania
  - Albert Einstein Cancer Center, Philadelphia, Pennsylvania
  - McGlinn Family Regional Cancer Center at Reading Hospital and Medical Center, Reading, Pennsylvania
  - Frank M. and Dorothea Henry Cancer Center at Geisinger Wyoming Valley Medical Center, Wilkes-Barre, Pennsylvania
  - Lankenau Cancer Center at Lankenau Hospital, Wynnewood, Pennsylvania
  - Hollings Cancer Center at Medical University of South Carolina, Charleston, South Carolina
  - Cancer Centers of the Carolinas - Faris Road, Greenville, South Carolina
  - CCOP - Greenville, Greenville, South Carolina
  - Cancer Centers of the Carolinas - Seneca, Seneca, South Carolina
  - Gibbs Regional Cancer Center at Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - Sanford Cancer Center at Sanford USD Medical Center, Sioux Falls, South Dakota
  - Christine LaGuardia Phillips Cancer Center at Wellmont Holston Valley Medical Center, Kingsport, Tennessee
  - Harrington Cancer Center, Amarillo, Texas
  - Texas Oncology, PA at Texas Cancer Center - Arlington South, Arlington, Texas
  - Texas Oncology, PA at Harris Center HEB, Bedford, Texas
  - Texas Oncology, PA at Texas Cancer Center - Denton South, Denton, Texas
  - Klabzuba Cancer Center at Harris Methodist Fort Worth Hospital, Fort Worth, Texas
  - M. D. Anderson Cancer Center at University of Texas, Houston, Texas
  - Longview Cancer Center, Longview, Texas
  - West Texas Cancer Center, Odessa, Texas
  - Cancer Care Centers of South Texas - Northeast, San Antonio, Texas
  - Texas Oncology, PA at Texas Cancer Center - Sherman, Sherman, Texas
  - Texas Oncology, PA at Texas Oncology Cancer Center Sugar Land, Sugar Land, Texas
  - Tyler Cancer Center, Tyler, Texas
  - Jon and Karen Huntsman Cancer Center at Intermountain Medical Center, Murray, Utah
  - Utah Valley Regional Medical Center - Provo, Provo, Utah
  - Utah Cancer Specialists at UCS Cancer Center, Salt Lake City, Utah
  - Dixie Regional Medical Center - East Campus, St. George, Utah
  - Fletcher Allen Health Care - University Health Center Campus, Burlington, Vermont
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - CCOP - Virginia Mason Research Center, Seattle, Washington
  - Cancer Care Northwest - Spokane South, Spokane, Washington
  - Theda Care Cancer Institute, Appleton, Wisconsin
  - Midelfort Clinic - Luther, Eau Claire, Wisconsin
  - Luther Midlelfort Hospital, Eau Claire, Wisconsin
  - Bellin Memorial Hospital, Green Bay, Wisconsin
  - St. Mary's Hospital Medical Center - Green Bay, Green Bay, Wisconsin
  - St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Gundersen Lutheran Center for Cancer and Blood, La Crosse, Wisconsin
  - Bay Area Cancer Care Center at Bay Area Medical Center, Marinette, Wisconsin
  - Medical College of Wisconsin Cancer Center, Milwaukee, Wisconsin
  - Veterans Affairs Medical Center - Milwaukee, Milwaukee, Wisconsin
  - D.N. Greenwald Center, Mukwonago, Wisconsin
  - All Saints Cancer Center at Wheaton Franciscan Healthcare, Racine, Wisconsin
  - Door County Cancer Center at Door County Memorial Hospital, Sturgeon Bay, Wisconsin
  - Waukesha Memorial Hospital Regional Cancer Center, Waukesha, Wisconsin
  - Riverview UW Cancer Center at Riverview Hospital, Wisconsin Rapids, Wisconsin
- Canada (6):
  - Tom Baker Cancer Centre - Calgary, Calgary, Alberta
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Princess Margaret Hospital, Toronto, Ontario
  - Hopital Notre-Dame du CHUM, Montreal, Quebec
  - Allan Blair Cancer Centre at Pasqua Hospital, Regina, Saskatchewan
  - Saskatoon Cancer Centre at the University of Saskatchewan, Saskatoon, Saskatchewan

REFERENCES:
- [Result] Bradley JD, Hu C, Komaki RR, Masters GA, Blumenschein GR, Schild SE, Bogart JA, Forster KM, Magliocco AM, Kavadi VS, Narayan S, Iyengar P, Robinson CG, Wynn RB, Koprowski CD, Olson MR, Meng J, Paulus R, Curran WJ Jr, Choy H. Long-Term Results of NRG Oncology RTOG 0617: Standard- Versus High-Dose Chemoradiotherapy With or Without Cetuximab for Unresectable Stage III Non-Small-Cell Lung Cancer. J Clin Oncol. 2020 Mar 1;38(7):706-714. doi: 10.1200/JCO.19.01162. Epub 2019 Dec 16. PMID 31841363
- [Derived] Chun SG, Hu C, Komaki RU, Timmerman RD, Schild SE, Bogart JA, Dobelbower MC, Bosch W, Kavadi VS, Narayan S, Iyengar P, Robinson C, Rothman J, Raben A, Augspurger ME, MacRae RM, Paulus R, Bradley JD. Long-Term Prospective Outcomes of Intensity Modulated Radiotherapy for Locally Advanced Lung Cancer: A Secondary Analysis of a Randomized Clinical Trial. JAMA Oncol. 2024 Aug 1;10(8):1111-1115. doi: 10.1001/jamaoncol.2024.1841. PMID 38935373
- [Derived] Zhang Z, Wang Z, Luo T, Yan M, Dekker A, De Ruysscher D, Traverso A, Wee L, Zhao L. Computed tomography and radiation dose images-based deep-learning model for predicting radiation pneumonitis in lung cancer patients after radiation therapy. Radiother Oncol. 2023 May;182:109581. doi: 10.1016/j.radonc.2023.109581. Epub 2023 Feb 25. PMID 36842666
- [Derived] McWilliam A, Abravan A, Banfill K, Faivre-Finn C, van Herk M. Demystifying the Results of RTOG 0617: Identification of Dose Sensitive Cardiac Subregions Associated With Overall Survival. J Thorac Oncol. 2023 May;18(5):599-607. doi: 10.1016/j.jtho.2023.01.085. Epub 2023 Feb 3. PMID 36738929
- [Derived] McKenzie E, Zhang S, Zakariaee R, Guthier CV, Hakimian B, Mirhadi A, Kamrava M, Padda SK, Lewis JH, Nikolova A, Mak RH, Atkins KM. Left Anterior Descending Coronary Artery Radiation Dose Association With All-Cause Mortality in NRG Oncology Trial RTOG 0617. Int J Radiat Oncol Biol Phys. 2023 Apr 1;115(5):1138-1143. doi: 10.1016/j.ijrobp.2022.11.033. Epub 2022 Nov 24. PMID 36436615
- [Derived] Movsas B, Hu C, Sloan J, Bradley J, Komaki R, Masters G, Kavadi V, Narayan S, Michalski J, Johnson DW, Koprowski C, Curran WJ Jr, Garces YI, Gaur R, Wynn RB, Schallenkamp J, Gelblum DY, MacRae RM, Paulus R, Choy H. Quality of Life Analysis of a Radiation Dose-Escalation Study of Patients With Non-Small-Cell Lung Cancer: A Secondary Analysis of the Radiation Therapy Oncology Group 0617 Randomized Clinical Trial. JAMA Oncol. 2016 Mar;2(3):359-67. doi: 10.1001/jamaoncol.2015.3969. PMID 26606200
- [Derived] Bradley JD, Paulus R, Komaki R, Masters G, Blumenschein G, Schild S, Bogart J, Hu C, Forster K, Magliocco A, Kavadi V, Garces YI, Narayan S, Iyengar P, Robinson C, Wynn RB, Koprowski C, Meng J, Beitler J, Gaur R, Curran W Jr, Choy H. Standard-dose versus high-dose conformal radiotherapy with concurrent and consolidation carboplatin plus paclitaxel with or without cetuximab for patients with stage IIIA or IIIB non-small-cell lung cancer (RTOG 0617): a randomised, two-by-two factorial phase 3 study. Lancet Oncol. 2015 Feb;16(2):187-99. doi: 10.1016/S1470-2045(14)71207-0. Epub 2015 Jan 16. PMID 25601342
- See also: Data Available: Select individual patient-level data from this trial can be requested from the NCTN/NCORP Data Archive. — https://nctn-data-archive.nci.nih.gov/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 60 Gy RT | 74 Gy RT | 60 Gy RT + Cetuximab | 74 Gy RT + Cetuximab
Started | 166 (Subjects with data available for the primary analysis are considered to have completed the study.) | 121 | 147 | 110
Completed | 151 | 107 | 137 | 100
Not Completed | 15 | 14 | 10 | 10
Not completed — Protocol Violation | 12 | 12 | 9 | 9
Not completed — Withdrawal by Subject | 3 | 2 | 1 | 1

BASELINE CHARACTERISTICS:
Population: All eligible patients who did not withdraw consent.
Groups:
- Total: Total of all reporting groups
Arm/Group | 60 Gy RT | 74 Gy RT | 60 Gy RT + Cetuximab | 74 Gy RT + Cetuximab | Total
Number analyzed (Participants) | 151 | 107 | 137 | 100 | 495
Age, Continuous [Median (Full Range); unit: years] | 64 [37 to 82] | 64 [41 to 82] | 64 [38 to 83] | 64 [44 to 83] | 64 [37 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54 | 39 | 60 | 47 | 200
  Male | 97 | 68 | 77 | 53 | 295

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: Survival time is defined as time from randomization to date of death from any cause and is estimated by the Kaplan-Meier method. Patients last known to be alive are censored at the date of last contact.
Time Frame: From randomization to last follow-up. Analysis occured after all patients were on study for 18 months. Maximum follow-up at time of analysis was 61.5 months.
Population: Eligible patients who did not withdraw consent; patients enrolled while high dose arms open to accrual are included in the RT comparison, patients enrolled while cetuximab arms open to accrual are included in the cetuximab comparison. See "Limitations and Caveats".
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Combined Patients Receiving 60 Gy RT: Combining patients from arms receiving 60 Gy radiation therapy (RT) (60 Gy RT and 60 Gy RT + Cetuximab)
- Combined Patients Receiving 74 Gy RT: Combining patients from arms receiving 74 Gy RT (74 Gy RT and 74 Gy RT + Cetuximab)
- Combined Patients Receiving Cetuximab: Combining patients from arms receiving Cetuximab (60 Gy RT + Cetuximab and 74 Gy RT + Cetuximab)
- Combined Patients From Arms Receiving No Cetuximab: Combining patients from arms receiving No Cetuximab (60 Gy RT and 74 Gy RT
Arm/Group | Combined Patients Receiving 60 Gy RT | Combined Patients Receiving 74 Gy RT | Combined Patients Receiving Cetuximab | Combined Patients From Arms Receiving No Cetuximab
Number analyzed (Participants) | 217 | 207 | 237 | 228
months | 28.7 [24.1 to 36.9] | 20.3 [17.7 to 25.0] | 25.0 [20.2 to 30.5] | 24.0 [19.8 to 28.6]
Statistical Analysis 1: Comparison: Combined Patients Receiving 60 Gy RT vs Combined Patients Receiving 74 Gy RT; The trial was a two-by-two factorial design with radiation therapy dose as one treatment factor and cetuximab as the other. A log-rank test for each factor at one-sided α of 0.0125 (α of 0.0250 for both factors to account for multiple comparisons) would yield power of 80% to detect an improvement in median survival from 17.1 to 24 months after 339 deaths were reported out of 500 patients. For RT analysis, the comparison was arms 1 & 3 vs arms 2 & 4; for cetuximab, arms 1 & 2 vs arms 3 & 4; Test type: Superiority or Other; p = 0.0042, Log Rank; Hazard Ratio (HR) = 1.38, 95% CI 2-sided [1.09 to 1.76] — Reference group = 60 gy
Statistical Analysis 2: Comparison: Combined Patients Receiving Cetuximab vs Combined Patients From Arms Receiving No Cetuximab; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.29, Log Rank; Hazard Ratio (HR) = 1.07, 95% CI 2-sided [0.84 to 1.35] — Reference level = cetuximab

2. Secondary Outcome: Progression-free Survival
Description: A failure for progression-free survival (PFS) is the first occurrence of local or regional progression, distant metastases, or death from any cause. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a nontarget lesion, or the appearance of new lesions. Time is measured from the date of randomization to the date of first failure. Patients without failure are censored at the date of last follow-up.
Time Frame: as for outcome 1
Population: Eligible patients who did not withdraw consent; patients enrolled while high dose arms open to accrual are included in the RT comparison, patients enrolled while cetuximab arms open to accrual are included in the cetuximab comparison.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Combined Patients Receiving 60 Gy RT: Combining patients from arms receiving 60 Gy RT (60 Gy RT and 60 Gy RT + Cetuximab)
Arm/Group | Combined Patients Receiving 60 Gy RT | Combined Patients Receiving 74 Gy RT | Combined Patients Receiving Cetuximab | Combined Patients From Arms Receiving No Cetuximab
Number analyzed (Participants) | 217 | 207 | 237 | 228
months | 11.8 [10.2 to 14.3] | 9.8 [8.8 to 11.6] | 10.8 [9.8 to 12.3] | 10.7 [9.3 to 13.2]
Statistical Analysis 1: Comparison: Combined Patients Receiving 60 Gy RT vs Combined Patients Receiving 74 Gy RT; Progression-free survival is estimated by the Kaplan-Meier method. Comparisons by RT level and by cetuximab assignment are performed separately and tested with a two-sided significance level of 0.05 for each comparison; Test type: Superiority or Other; p = 0.12, Log Rank; Hazard Ratio (HR) = 1.19, 95% CI 2-sided [0.95 to 1.47] — Reference level = 60 Gy
Statistical Analysis 2: Comparison: Combined Patients Receiving Cetuximab vs Combined Patients From Arms Receiving No Cetuximab; Progression-free survival is estimated by the Kaplan-Meier method. Comparisons by RT level and by cetuximab assignment are performed separately and tested with a two-sided significance level of 0.05; Test type: Superiority or Other; p = 0.89, Log Rank; Hazard Ratio (HR) = 0.99, 95% CI 2-sided [0.80 to 1.22] — Reference level = cetuximab

3. Secondary Outcome: Local-regional Failure (Reported as Two-year Estimates)
Description: A failure for local-regional failure is the first occurrence of local or regional progression. Time is measured from the date of randomization to the date of first failure. Patients alive without local or regional failure at the time of last follow-up are censored. Patients who died without local or regional failure are considered as having competing risk at the time of death. Local-regional failure was estimated by the cumulative incidence method and 2 year estimates are reported.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Combined Patients Receiving 60 Gy RT | Combined Patients Receiving 74 Gy RT | Combined Patients Receiving Cetuximab | Combined Patients From Arms Receiving No Cetuximab
Number analyzed (Participants) | 217 | 207 | 237 | 228
percentage of participants | 42.3 [35.7 to 49.0] | 48.4 [41.5 to 55.3] | 47.1 [40.6 to 53.6] | 40.7 [34.2 to 47.3]
Statistical Analysis 1: Comparison: Combined Patients Receiving 60 Gy RT vs Combined Patients Receiving 74 Gy RT; Local-regional failure was estimated by the cumulative incidence method. Comparisons by RT level and by cetuximab assignment are performed separately and tested with a two-sided significance level of 0.05 for each comparison; Test type: Superiority or Other; p = 0.24, Gray's test; Hazard Ratio (HR) = 1.17, 95% CI 2-sided [0.89 to 1.53] — Reference level = 60 Gy
Statistical Analysis 2: Comparison: Combined Patients Receiving Cetuximab vs Combined Patients From Arms Receiving No Cetuximab; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.22, Gray's test; Hazard Ratio (HR) = 0.84, 95% CI 2-sided [0.64 to 1.10] — Reference level = cetuximab

4. Secondary Outcome: Percentage of Participants With Grade 3-5 Esophagitis and Pneumonitis Adverse Events as Assessed by NCI Common Toxicity Criteria for Adverse Effects (CTCAE) v3.0
Description: Treatment-related esophagitis and pneumonitis were assessed graded using the CTCAE v3.0. Comparisons are only made between radiation therapy dosing levels because the cetuximab regimen was known to be safe in combination with radiation therapy.
Time Frame: as for outcome 1
Population: All eligible patients enrolled while the high dose arms were open, who did not withdraw consent.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Combined Patients Receiving 60 Gy RT | Combined Patients Receiving 74 Gy RT
Number analyzed (Participants) | 217 | 207
percentage of participants
  Esophagitis | 7.4 [4.3 to 11.7] | 20.8 [15.5 to 26.9]
  Pneumonitis | 6.9 [3.5 to 10.3] | 4.3 [2.0 to 8.1]
Statistical Analysis 1: Comparison: Combined Patients Receiving 60 Gy RT vs Combined Patients Receiving 74 Gy RT; Esophagitis: Only those toxicities reported as possibly, probably, or definitely related to treatment were considered. The worst grade of esophagitis and the worst grade of pneumonitis at any time were classified by binary groupings of < grade 3 and >= grade 3. Comparisons were made using a two-sided chi-square test with a significance level of 0.05; Test type: Superiority or Other; p < 0.0001, Chi-squared
Statistical Analysis 2: Comparison: Combined Patients Receiving 60 Gy RT vs Combined Patients Receiving 74 Gy RT; PNEUMONITIS: Only those toxicities reported as possibly, probably, or definitely related to treatment were considered. The worst grade of esophagitis and the worst grade of pneumonitis at any time were classified by binary groupings of < grade 3 and >= grade 3. Comparisons were made using a two-sided chi-square test with a significance level of 0.05; Test type: Superiority or Other; p = 0.2533, Chi-squared

5. Secondary Outcome: Percentage of Participants With Other Grade 3-5 Adverse Events as Assessed by NCI CTCAE v3.0
Description: Treatment-related adverse events other than esophagitis and pneumonitis were assessed graded using the CTCAE v3.0. Comparisons are only made between radiation therapy dosing levels because the cetuximab regimen was known to be safe in combination with radiation therapy.
Time Frame: as for outcome 1
Population: All eligible patients enrolled while the high dose arms were open, who did not withdraw consent.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Combined Patients Receiving 60 Gy RT | Combined Patients Receiving 74 Gy RT
Number analyzed (Participants) | 217 | 207
percentage of participants | 75.1 [68.8 to 80.7] | 77.8 [71.5 to 83.3]
Statistical Analysis 1: Comparison: Combined Patients Receiving 60 Gy RT vs Combined Patients Receiving 74 Gy RT; Only those toxicities reported as possibly, probably, or definitely related to treatment were considered. The worst grade of of toxicity at any time was classified by a binary grouping of < grade 3 and >= grade 3. Comparisons were made using a two-sided chi-square test; Test type: Superiority or Other; p = 0.52, Chi-squared

6. Secondary Outcome: Death During or Within 30 Days of Discontinuation of Protocol Treatment
Description: Deaths regardless of cause and occuring during or within 30 days of discontinuation of protocol treatment were evaluated.
Time Frame: From start of protocol treatment to 24 months.
Population: Eligible patients who started study treatment and did not withdraw consent.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 60 Gy RT | 74 Gy RT | 60 Gy RT + Cetuximab | 74 Gy RT + Cetuximab
Number analyzed (Participants) | 148 | 106 | 136 | 98
percentage of participants | 2 [0 to 4.3] | 3.8 [0.1 to 7.4] | 8.8 [4.1 to 13.6] | 4.1 [0.2 to 8.0]

7. Secondary Outcome: Percentage of Patients With Decline From Baseline to 3 Months in the Lung Cancer Subscale (LCS) of the Functional Assessment of the Cancer Therapy Trial Outcome Index (FACT-TOI).
Description: A decline of 2 points in the LCS from baseline to 3 months was considered a clinically meaningful change indicating a decline in quality of life. Comparisons are only made between radiation therapy dosing levels because the cetuximab regimen was known to be safe in combination with radiation therapy.
Time Frame: At baseline and 3 months.
Population: Eligible patients who enrolled while the high dose arms were open, had baseline and 3 month assessments, and did not withdraw consent.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Combined Patients Receiving 60 Gy RT | Combined Patients Receiving 74 Gy RT
Number analyzed (Participants) | 107 | 109
percentage of participants | 29.9 [21.4 to 39.5] | 45.0 [35.4 to 54.8]
Statistical Analysis 1: Comparison: Combined Patients Receiving 60 Gy RT vs Combined Patients Receiving 74 Gy RT; FACT-TOI-LCS was assessed and changes from baseline to 3 months calculated and grouped using a 2 point decline as the threshold. Comparisons of decline vs no decline by RT level were from a Cochran-Mantel-Haenszel test and controlling for cetuximab assignment using a two-side significance level of 0.05; Test type: Superiority or Other; p = 0.0233, Cochran-Mantel-Haenszel

8. Secondary Outcome: Patient-reported Swallowing Score (Area Under the Curve)
Description: Patients completed a swallowing diary prior to the start of treatment and then daily during treatment. Patients recorded a score to indicate problems with swallowing on that day (1-None, 2-Mild soreness only, 3-Can swallow solids with some difficulty, 4-Cannot swallow solids, 5-Cannot swallow liquids). These scores were then plotted across time and the area under the curve from baseline until the end of week 6 was calculated. A lower area under the curve indicates better swallowing ability. Comparisons are only made between radiation therapy dosing levels because the cetuximab regimen was known to be safe in combination with radiation therapy.
Time Frame: From randomization to 6 weeks after start of radiation therapy (6-10 weeks from randomization)
Population: Eligible patients enrolled while the high radiation therapy dose arms were open to accrual and who had at least 15 diary entries including one prior to start of radiation therapy and one during sixth week from start of radiation therapy.
Measure: Median (Inter-Quartile Range); unit: Area under curve (score * days)
Arm/Group | Combined Patients Receiving 60 Gy RT | Combined Patients Receiving 74 Gy RT
Number analyzed (Participants) | 135 | 125
Area under curve (score * days) | 79.5 [59.5 to 99.0] | 78.0 [55.5 to 97.0]
Statistical Analysis 1: Comparison: Combined Patients Receiving 60 Gy RT vs Combined Patients Receiving 74 Gy RT; Test type: Superiority; p = 0.92, t-test, 2 sided; Two-sided significance level = 0.05

9. Secondary Outcome: EuroQoL (EQ5D) Visual Analog Scale (VAS) Through One Year (Area Under the Curve)
Description: The visual analogue scale is a self-assessment of current health state, measured on a 20-cm scale ranging from 0 for the worst imaginable health state to 100 for best imaginable health state, marked at 10-point intervals. The area under the curve of each subject's EQ5D visual analog scale (VAS) response trajectory within 1 year was calculated. The EQ5D VAS utility was normalized by the baseline score. The trajectory included all available time points through one year. If a subject died within one year, the EQ5D VAS was reduced to 0 at the time of death. If subject was censored within one year, the EQ5D utility curve was truncated at the time of censoring. The scores were plotted across time and the area under the curve was calculated. A greater area under the curve indicates a better health state. Comparisons are only made between radiation therapy dosing levels because the cetuximab regimen was known to be safe in combination with radiation
Time Frame: From randomization to one year
Population: Eligible patients enrolled while the high radiation therapy dose arms were open to accrual, started treatment, and had baseline and at least one follow-up EQ5D VAS.
Measure: Median (Inter-Quartile Range); unit: Score on a scale * months
Arm/Group | Combined Patients Receiving 60 Gy RT | Combined Patients Receiving 74 Gy RT
Number analyzed (Participants) | 135 | 118
Score on a scale * months | 279.5 [40.4 to 1852.4] | 265.4 [55.9 to 76.9]
Statistical Analysis 1: Comparison: Combined Patients Receiving 60 Gy RT vs Combined Patients Receiving 74 Gy RT; Test type: Superiority; p = 0.19, t-test, 2 sided; Two-sided significance level = 0.05

10. Secondary Outcome: Overall Survival and Local-regional Failure by Epithelial Growth Factor Receptor (EGFR) Group
Description: EGFR is a protein that is present on the surface of both normal cells and cancer cancer cells. EGFR H-Score is a measure of staining intensity ranging from 0 to 300 where a higher value indicates greater intensity of EGFR. Available tumor samples were evaluated for EGFR and given an H-Score. Patients were divided into two groups based on H-Score values dichotomized at 200. All event times are time from randomization to date of event or censoring. A survival event is death from any cause, patients without events are censored at the date of last contact, and survival rates are estimated by Kaplan-Meier method. A local-regional event is the first development of progressive disease locally or regionally, patients who do not have an event are censored at the date of death or last contact, and event rates are estimated by cumulative incidence. Two-year rates are reported.
Time Frame: as for outcome 1
Population: Eligible patients with EGFR H-Score
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | EGFR H-Score < 200 | EGFR H-Score >= 200
Number analyzed (Participants) | 111 | 109
percentage of participants
  Two-year Survival rate | 51.7 [41.9 to 60.6] | 52.8 [42.9 to 61.7]
  Two-year Local-regional Failure rate | 37.4 [28.3 to 46.6] | 47.2 [37.7 to 56.7]
Statistical Analysis 1: Comparison: EGFR H-Score < 200 vs EGFR H-Score >= 200; Univariate model of overall survival by EGFR group; Test type: Superiority; p = 0.78, Regression, Cox; Hazard Ratio (HR) = 0.95, 95% CI 2-sided [0.68 to 1.33] — Reference level = EGFR H-Score < 200
Statistical Analysis 2: Comparison: EGFR H-Score < 200 vs EGFR H-Score >= 200; Univariate model of time to local-regional failure by EGFR group; Test type: Superiority; p = 0.61, Regression, Cox; Hazard Ratio (HR) = 1.11, 95% CI 2-sided [0.74 to 1.65] — Reference level = EGFR H-Score < 200

11. Secondary Outcome: Percentage of Patients With Grade 3+ Adverse Events by Epithelial Growth Factor Receptor (EGFR) Group
Description: EGFR is a protein that is present on the surface of both normal cells and cancer cancer cells. EGFR H-Score is a measure of staining intensity ranging from 0 to 300 where a higher value indicates greater intensity of EGFR. Available tumor samples were evaluated for EGFR and given an H-Score. Patients were divided into two groups based on H-Score values dichotomized at 200. Worst toxicity as determined by adverse events was used as a measure of a patient's quality of life (QOL). Adverse events were graded using the Common Terminology Criteria for Adverse Events (CTCAE) v3.0. Grade refers to the severity of the AE. The CTCAE v3.0 assigns Grades 1 through 5 with unique clinical descriptions of severity for each AE based on this general guideline: Grade 1 Mild, Grade 2 Moderate, Grade 3 Severe, Grade 4 Life-threatening or disabling, Grade 5 Death related to AE. Highest grade (worst) adverse event (AE) per subject was counted.
Time Frame: as for outcome 1
Population: Eligible patients with EGFR H-Score
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | EGFR H-Score < 200 | EGFR H-Score >= 200
Number analyzed (Participants) | 111 | 109
percentage of participants | 72.1 [63.7 to 80.4] | 85.3 [78.7 to 92.0]
Statistical Analysis 1: Comparison: EGFR H-Score < 200 vs EGFR H-Score >= 200; Test type: Superiority; p = 0.02, Chi-squared — Two-sided significance level = 0.05

12. Secondary Outcome: Prognostic and Predictive Effects of Gross Tumor Volume (GTV) on Overall Survival
Description: Gross tumor volume (GTV) is defined as the combined volume (cubic centimeters) of the primary tumor and clinically positive lymph nodes seen either on the planning computed tomography (CT) scan or the pretreatment positron emission tomography (PET) scan. Survival time is defined as time from randomization to date of death from any cause and is estimated by the Kaplan-Meier method. Patients last known to be alive are censored at the date of last contact. GTV was evaluated as a continuous variable therefore overall survival time is not summarized by GTV. "Prognostic" refers to the main effect and "predictive" refers to the interaction between GTV and treatment arm.
Time Frame: as for outcome 1
Population: Eligible patients with GTV data
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | All Patients
Number analyzed (Participants) | 356
months | 25.0 [20.6 to 28.6]
Statistical Analysis 1: Comparison: All Patients; Univariate model with GTV as a continuous variable; Test type: Other; p = 0.06, Regression, Cox — Two-sided significance level = 0.05; Cox Proportional Hazard = 1.001, 95% CI 2-sided [1.000 to 1.002] — Corresponding to a one unit increase in GTV
Statistical Analysis 2: Comparison: All Patients; Multivariate model with GTV as a continuous variable, adjusting for planned radiation therapy dose group (60 Gy or 74 Gy) and the interaction of GTV and planned dose; Test type: Superiority; p = 0.78, Regression, Cox — Two-sided significance level = 0.05; Hazard Ratio (HR) = 1.001, 95% CI 2-sided [0.997 to 1.004] — Corresponding to a one unit increase in GTV; P-Value for the interaction of GTV and planned dose = 0.77

13. Secondary Outcome: Prognostic Value of Pre-treatment Standardized Uptake Value (SUV) of Positron Emission Tomography (PET) Scan in Predicting Survival, Distant Metastasis, and Local-regional Failure
Description: Standardized uptake value (SUV) is a simple way of determining activity in PET imaging. It is a mathematically derived ratio of tissue radioactivity concentration at a point in time and the injected dose of radioactivity per kilogram of the patient's body weight. All event times are time from randomization to date of event or censoring. A survival event is death from any cause, patients without events are censored at the date of last contact, and survival rates are estimated by Kaplan-Meier method. Local-regional and distant metastasis events are the first development of progressive disease locally/regionally or distant metastasis, respectively, patients who do not have an event are censored at the date of death or last contact, and event rates are estimated by cumulative incidence. Two-year rates are presented. PET SUV was evaluated as a continuous variable therefore the outcome variables are not summarized by PET SUV.
Time Frame: as for outcome 1
Population: Eligible patients with PET SUV data at baseline.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | All Patients
Number analyzed (Participants) | 444
percentage of participants
  Overall Survival | 50.5 [45.7 to 55.2]
  Time to Distant Metastasis | 46.7 [41.9 to 51.3]
  Time to Local-Regional Failure | 43.7 [38.9 to 48.3]
Statistical Analysis 1: Comparison: All Patients; Univariate model of overall survival time by PET SUV as a continuous variable; Test type: Superiority; p = 0.94, Regression, Cox; Cox Proportional Hazard = 1.00, 95% CI 2-sided [0.98 to 1.02] — Corresponding to a one unit increase in SUV
Statistical Analysis 2: Comparison: All Patients; Univariate model of time to local-regional failure by PET SUV as a continuous variable; Test type: Superiority; p = 0.72, Regression, Cox; Cox Proportional Hazard = 1.00, 95% CI 2-sided [0.98 to 1.02] — Corresponding to a one unit increase in SUV
Statistical Analysis 3: Comparison: All Patients; Univariate model of time to distant metastasis by PET SUV as a continuous variable; Test type: Superiority; p = 0.79, Regression, Cox; Cox Proportional Hazard = 1.00, 95% CI 2-sided [0.98 to 1.02] — Corresponding to a one unit increase in SUV

ADVERSE EVENTS:
Description: Eligible patients with adverse event data are included. Patients experiencing more than one of a given adverse event are counted only once for that adverse event.
Arm/Group | 60 Gy RT | 74 Gy RT | 60 Gy RT + Cetuximab | 74 Gy RT + Cetuximab
Serious Adverse Events (participants affected / at risk) | 60/149 | 49/104 | 84/134 | 57/97
Other Adverse Events (participants affected / at risk) | 145/149 | 102/104 | 129/134 | 95/97
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 60 Gy RT (N=149) | 74 Gy RT (N=104) | 60 Gy RT + Cetuximab (N=134) | 74 Gy RT + Cetuximab (N=97)
Blood disorder (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 3 | 4 | 8 | 3
Hemoglobin decreased (Blood and lymphatic system disorders) | 10 | 7 | 8 | 7
Hemolysis (Blood and lymphatic system disorders) | 1 | 0 | 2 | 0
Arrhythmia (Cardiac disorders) | 0 | 1 | 2 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 4 | 5 | 1
Atrial flutter (Cardiac disorders) | 0 | 0 | 1 | 1
Atrial tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0
Cardiac disorder (Cardiac disorders) | 1 | 2 | 1 | 2
Cardiac pain (Cardiac disorders) | 1 | 0 | 0 | 0
Cardiopulmonary arrest (Cardiac disorders) | 2 | 0 | 0 | 0
Myocardial ischemia (Cardiac disorders) | 1 | 0 | 1 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 1 | 0
Pericardial effusion (Cardiac disorders) | 1 | 1 | 0 | 1
Pericarditis (Cardiac disorders) | 1 | 0 | 0 | 0
Premature ventricular contractions (Cardiac disorders) | 0 | 1 | 0 | 0
Restrictive cardiomyopathy (Cardiac disorders) | 0 | 0 | 0 | 1
Sinus tachycardia (Cardiac disorders) | 1 | 1 | 0 | 2
Supraventricular tachycardia (Cardiac disorders) | 0 | 1 | 0 | 1
Ventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 1 | 0 | 1 | 0
Dry eye syndrome (Eye disorders) | 0 | 0 | 1 | 0
Watering eyes (Eye disorders) | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 5 | 2
Acquired tracheo-esophageal fistula (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Colonic fistula (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Colonic perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 2 | 6 | 0
Diarrhea (Gastrointestinal disorders) | 4 | 1 | 4 | 3
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Duodenal hemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Duodenal ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 2 | 3 | 0
Dysphagia (Gastrointestinal disorders) | 3 | 11 | 7 | 9
Esophageal hemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Esophageal mucositis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Esophageal pain (Gastrointestinal disorders) | 1 | 5 | 1 | 3
Esophageal perforation (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Esophageal stenosis (Gastrointestinal disorders) | 1 | 2 | 0 | 3
Esophageal ulcer (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Esophagitis (Gastrointestinal disorders) | 6 | 14 | 10 | 7
Gastric hemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastrointestinal disorder (Gastrointestinal disorders) | 1 | 0 | 0 | 3
Gastrointestinal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Ileal perforation (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Mucositis oral (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Nausea (Gastrointestinal disorders) | 7 | 2 | 10 | 7
Rectal hemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Vomiting (Gastrointestinal disorders) | 3 | 0 | 6 | 5
Chest pain (General disorders) | 2 | 4 | 1 | 0
Chills (General disorders) | 0 | 0 | 4 | 0
Death (General disorders) | 0 | 0 | 2 | 1
Disease progression (General disorders) | 0 | 2 | 1 | 0
Edema limbs (General disorders) | 1 | 0 | 0 | 1
Fatigue (General disorders) | 6 | 9 | 11 | 12
Fever (General disorders) | 5 | 7 | 9 | 1
Flu-like symptoms (General disorders) | 0 | 0 | 1 | 0
Gait abnormal (General disorders) | 0 | 0 | 1 | 0
General symptom (General disorders) | 1 | 0 | 1 | 0
Ill-defined disorder (General disorders) | 0 | 0 | 1 | 1
Pain [other] (General disorders) | 2 | 1 | 1 | 0
Sudden death (General disorders) | 0 | 1 | 2 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Cytokine release syndrome (Immune system disorders) | 0 | 0 | 1 | 0
Hypersensitivity (Immune system disorders) | 1 | 2 | 6 | 4
Appendicitis perforated (Infections and infestations) | 0 | 0 | 0 | 1
Bladder infection [with unknown ANC] (Infections and infestations) | 0 | 0 | 0 | 1
Bone infection [with normal or Grade 1-2 ANC] (Infections and infestations) | 0 | 0 | 1 | 0
Bronchitis [with Grade 3-4 ANC] (Infections and infestations) | 0 | 0 | 1 | 0
Bronchitis [with normal or Grade 1-2 ANC] (Infections and infestations) | 1 | 0 | 2 | 0
Bronchitis [with unknown ANC] (Infections and infestations) | 0 | 1 | 0 | 0
Catheter related infection [with Grade 3-4 ANC] (Infections and infestations) | 0 | 0 | 1 | 0
Catheter related infection [with normal or Grade 1-2 ANC] (Infections and infestations) | 0 | 0 | 1 | 0
Catheter related infection [with unknown ANC] (Infections and infestations) | 0 | 0 | 1 | 0
Colitis, infectious (e.g., Clostridium difficile) (Infections and infestations) | 0 | 0 | 0 | 1
Device related infection [with unknown ANC] (Infections and infestations) | 0 | 0 | 1 | 0
Endocarditis infective [with normal or Grade 1-2 ANC] (Infections and infestations) | 0 | 0 | 1 | 0
Endocarditis infective [with unknown ANC] (Infections and infestations) | 0 | 0 | 1 | 0
Gingival infection [with Grade 3-4 ANC] (Infections and infestations) | 0 | 0 | 0 | 1
Gingival infection [with unknown ANC] (Infections and infestations) | 1 | 0 | 0 | 0
Infection [other] (Infections and infestations) | 0 | 3 | 1 | 1
Infectious colitis [with unknown ANC] (Infections and infestations) | 0 | 0 | 0 | 1
Opportunistic infection (Infections and infestations) | 0 | 1 | 0 | 0
Penile infection [with Grade 3-4 ANC] (Infections and infestations) | 0 | 0 | 0 | 1
Peritoneal infection [with normal or Grade 1-2 ANC] (Infections and infestations) | 0 | 0 | 1 | 0
Pleural infection [with normal or Grade 1-2 ANC] (Infections and infestations) | 0 | 1 | 0 | 0
Pneumonia [with Grade 3-4 ANC] (Infections and infestations) | 3 | 1 | 2 | 1
Pneumonia [with normal or Grade 1-2 ANC] (Infections and infestations) | 7 | 6 | 5 | 1
Pneumonia [with unknown ANC] (Infections and infestations) | 1 | 4 | 5 | 3
Sepsis [with Grade 3-4 ANC] (Infections and infestations) | 0 | 0 | 1 | 0
Sepsis [with normal or Grade 1-2 ANC] (Infections and infestations) | 0 | 0 | 1 | 2
Sepsis [with unknown ANC] (Infections and infestations) | 0 | 0 | 2 | 0
Skin infection [with Grade 3-4 ANC] (Infections and infestations) | 0 | 0 | 0 | 1
Skin infection [with normal or Grade 1-2 ANC] (Infections and infestations) | 0 | 0 | 0 | 1
Soft tissue infection [with normal or Grade 1-2 ANC] (Infections and infestations) | 0 | 1 | 0 | 0
Upper respiratory infection [with normal or Grade 1-2 ANC] (Infections and infestations) | 0 | 1 | 1 | 0
Urinary tract infection [with Grade 3-4 ANC] (Infections and infestations) | 0 | 0 | 1 | 0
Urinary tract infection [with normal or Grade 1-2 ANC] (Infections and infestations) | 1 | 1 | 0 | 0
Urinary tract infection [with unknown ANC] (Infections and infestations) | 1 | 0 | 0 | 0
Wound infection [with Grade 3-4 ANC] (Infections and infestations) | 0 | 0 | 0 | 1
Wound infection [with normal or Grade 1-2 ANC] (Infections and infestations) | 0 | 1 | 0 | 0
Dermatitis radiation (Injury, poisoning and procedural complications) | 2 | 1 | 1 | 3
Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Intraoperative musculoskeletal injury - Joint (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Radiation recall reaction (dermatologic) (Injury, poisoning and procedural complications) | 1 | 1 | 2 | 1
Thermal burn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Vascular access complication (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 1
Activated partial thromboplastin time prolonged (Investigations) | 0 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0 | 1
Alkaline phosphatase increased (Investigations) | 0 | 1 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 0 | 1
CD4 lymphocytes decreased (Investigations) | 0 | 0 | 1 | 0
Carbon monoxide diffusing capacity decreased (Investigations) | 0 | 0 | 0 | 1
Creatinine increased (Investigations) | 1 | 0 | 1 | 0
Forced expiratory volume decreased (Investigations) | 0 | 0 | 0 | 1
INR increased (Investigations) | 0 | 0 | 0 | 1
Laboratory test abnormal (Investigations) | 0 | 0 | 2 | 1
Leukopenia (Investigations) | 6 | 8 | 13 | 8
Lymphopenia (Investigations) | 3 | 5 | 6 | 2
Neutrophil count decreased (Investigations) | 10 | 13 | 17 | 13
Platelet count decreased (Investigations) | 6 | 3 | 5 | 9
Weight loss (Investigations) | 4 | 8 | 8 | 5
Anorexia (Metabolism and nutrition disorders) | 2 | 3 | 8 | 6
Dehydration (Metabolism and nutrition disorders) | 11 | 7 | 23 | 14
Glucose intolerance (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 2 | 2 | 2 | 3
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 | 1 | 2 | 4
Hypocalcemia (Metabolism and nutrition disorders) | 2 | 1 | 3 | 2
Hypoglycemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 3 | 2 | 5 | 6
Hypomagnesemia (Metabolism and nutrition disorders) | 1 | 2 | 6 | 2
Hyponatremia (Metabolism and nutrition disorders) | 2 | 2 | 1 | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2 | 2
Muscle weakness (Musculoskeletal and connective tissue disorders) | 2 | 1 | 1 | 2
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0
Soft tissue necrosis lower limb (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Ataxia (Nervous system disorders) | 1 | 0 | 1 | 1
Cognitive disturbance (Nervous system disorders) | 0 | 0 | 1 | 0
Depressed level of consciousness (Nervous system disorders) | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 2 | 0 | 1 | 1
Extrapyramidal disorder (Nervous system disorders) | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 0 | 1 | 1
Ischemia cerebrovascular (Nervous system disorders) | 0 | 1 | 3 | 2
Leukoencephalopathy (Nervous system disorders) | 0 | 0 | 1 | 0
Peripheral motor neuropathy (Nervous system disorders) | 1 | 0 | 1 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0 | 1 | 3
Syncope (Nervous system disorders) | 1 | 0 | 4 | 0
Syncope vasovagal (Nervous system disorders) | 0 | 0 | 1 | 0
Taste alteration (Nervous system disorders) | 0 | 0 | 1 | 1
Agitation (Psychiatric disorders) | 0 | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 3 | 0 | 0 | 1
Confusion (Psychiatric disorders) | 1 | 0 | 3 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 1 | 0 | 1 | 0
Hemoglobinuria (Renal and urinary disorders) | 0 | 0 | 1 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 1 | 1
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 1
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 1
Bronchial fistula (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 3 | 3 | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 18 | 12 | 17 | 10
Hemorrhage nasal (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 5 | 0 | 2 | 4
Pharyngeal examination abnormal (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 0 | 2
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 4 | 5 | 11 | 5
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 3 | 1
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 3 | 1
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 3 | 3 | 5 | 3
Respiratory tract hemorrhage (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1 | 0
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 2 | 1
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 9 | 3
Alopecia (Skin and subcutaneous tissue disorders) | 2 | 0 | 3 | 1
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 4 | 1
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Nail disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Photosensitivity (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1
Rash desquamating (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 1
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Hemorrhage (Vascular disorders) | 0 | 1 | 1 | 0
Hypotension (Vascular disorders) | 4 | 1 | 8 | 3
Thrombosis (Vascular disorders) | 5 | 6 | 4 | 9
Vascular disorder (Vascular disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 60 Gy RT (N=149) | 74 Gy RT (N=104) | 60 Gy RT + Cetuximab (N=134) | 74 Gy RT + Cetuximab (N=97)
Hemoglobin decreased (Blood and lymphatic system disorders) | 90 | 63 | 69 | 58
Sinus tachycardia (Cardiac disorders) | 3 | 5 | 6 | 8
Vision blurred (Eye disorders) | 4 | 3 | 3 | 6
Abdominal pain (Gastrointestinal disorders) | 6 | 5 | 11 | 8
Constipation (Gastrointestinal disorders) | 55 | 34 | 45 | 48
Diarrhea (Gastrointestinal disorders) | 37 | 15 | 45 | 34
Dry mouth (Gastrointestinal disorders) | 7 | 2 | 2 | 5
Dyspepsia (Gastrointestinal disorders) | 21 | 12 | 36 | 23
Dysphagia (Gastrointestinal disorders) | 72 | 47 | 73 | 57
Ear, nose and throat examination abnormal (Gastrointestinal disorders) | 7 | 5 | 7 | 4
Esophageal pain (Gastrointestinal disorders) | 11 | 18 | 12 | 11
Esophageal stenosis (Gastrointestinal disorders) | 3 | 7 | 2 | 7
Esophagitis (Gastrointestinal disorders) | 65 | 51 | 56 | 52
Mucositis oral (Gastrointestinal disorders) | 15 | 8 | 29 | 17
Nausea (Gastrointestinal disorders) | 68 | 50 | 65 | 53
Vomiting (Gastrointestinal disorders) | 29 | 19 | 41 | 27
Chest pain (General disorders) | 27 | 19 | 19 | 20
Chills (General disorders) | 7 | 4 | 11 | 11
Edema limbs (General disorders) | 14 | 10 | 10 | 9
Fatigue (General disorders) | 112 | 77 | 97 | 83
Fever (General disorders) | 21 | 20 | 25 | 28
Pain [NOS] (General disorders) | 6 | 2 | 6 | 6
Pain [other] (General disorders) | 13 | 12 | 17 | 15
Hypersensitivity (Immune system disorders) | 8 | 8 | 13 | 12
Infection [other] (Infections and infestations) | 5 | 7 | 5 | 3
Pneumonia [with normal or Grade 1-2 ANC] (Infections and infestations) | 10 | 3 | 2 | 7
Dermatitis radiation (Injury, poisoning and procedural complications) | 44 | 36 | 45 | 39
Radiation recall reaction (dermatologic) (Injury, poisoning and procedural complications) | 16 | 19 | 33 | 18
Alanine aminotransferase increased (Investigations) | 22 | 14 | 17 | 20
Alkaline phosphatase increased (Investigations) | 14 | 10 | 17 | 12
Aspartate aminotransferase increased (Investigations) | 17 | 9 | 16 | 20
Creatinine increased (Investigations) | 12 | 8 | 7 | 7
Hyperbilirubinemia (Investigations) | 4 | 3 | 7 | 4
Laboratory test abnormal (Investigations) | 12 | 2 | 14 | 5
Leukopenia (Investigations) | 79 | 58 | 67 | 55
Lymphopenia (Investigations) | 44 | 28 | 33 | 19
Neutrophil count decreased (Investigations) | 58 | 41 | 69 | 58
Platelet count decreased (Investigations) | 60 | 43 | 48 | 41
Weight loss (Investigations) | 60 | 50 | 68 | 56
Anorexia (Metabolism and nutrition disorders) | 43 | 36 | 48 | 49
Dehydration (Metabolism and nutrition disorders) | 19 | 8 | 29 | 19
Hypercalcemia (Metabolism and nutrition disorders) | 5 | 4 | 9 | 4
Hyperglycemia (Metabolism and nutrition disorders) | 42 | 25 | 43 | 34
Hyperkalemia (Metabolism and nutrition disorders) | 9 | 7 | 5 | 7
Hypernatremia (Metabolism and nutrition disorders) | 3 | 2 | 7 | 3
Hypoalbuminemia (Metabolism and nutrition disorders) | 27 | 20 | 33 | 29
Hypocalcemia (Metabolism and nutrition disorders) | 24 | 16 | 29 | 20
Hypokalemia (Metabolism and nutrition disorders) | 23 | 17 | 33 | 26
Hypomagnesemia (Metabolism and nutrition disorders) | 17 | 12 | 67 | 49
Hyponatremia (Metabolism and nutrition disorders) | 32 | 26 | 36 | 27
Back pain (Musculoskeletal and connective tissue disorders) | 15 | 11 | 16 | 7
Chest wall pain (Musculoskeletal and connective tissue disorders) | 12 | 6 | 12 | 9
Joint pain (Musculoskeletal and connective tissue disorders) | 28 | 11 | 11 | 10
Muscle weakness (Musculoskeletal and connective tissue disorders) | 12 | 6 | 6 | 14
Myalgia (Musculoskeletal and connective tissue disorders) | 21 | 15 | 12 | 6
Pain in extremity (Musculoskeletal and connective tissue disorders) | 12 | 2 | 13 | 9
Dizziness (Nervous system disorders) | 23 | 19 | 21 | 10
Headache (Nervous system disorders) | 31 | 20 | 37 | 26
Neurological disorder NOS (Nervous system disorders) | 8 | 1 | 4 | 4
Peripheral motor neuropathy (Nervous system disorders) | 15 | 6 | 7 | 4
Peripheral sensory neuropathy (Nervous system disorders) | 60 | 42 | 51 | 40
Taste alteration (Nervous system disorders) | 10 | 10 | 20 | 13
Anxiety (Psychiatric disorders) | 18 | 5 | 11 | 7
Depression (Psychiatric disorders) | 13 | 8 | 6 | 9
Insomnia (Psychiatric disorders) | 22 | 13 | 16 | 19
Urinary frequency (Renal and urinary disorders) | 4 | 4 | 3 | 5
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 6 | 2 | 4 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 83 | 55 | 72 | 52
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 82 | 59 | 62 | 51
Hemorrhage nasal (Respiratory, thoracic and mediastinal disorders) | 12 | 11 | 18 | 11
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 10 | 5 | 5 | 6
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 11 | 7 | 7 | 7
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 11 | 8 | 7 | 7
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 29 | 13 | 20 | 15
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 14 | 7 | 13 | 6
Pulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 7 | 2 | 1 | 9
Respiratory tract hemorrhage (Respiratory, thoracic and mediastinal disorders) | 7 | 5 | 7 | 3
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 13 | 9 | 8 | 11
Acne (Skin and subcutaneous tissue disorders) | 11 | 7 | 105 | 68
Alopecia (Skin and subcutaneous tissue disorders) | 46 | 33 | 27 | 31
Dry skin (Skin and subcutaneous tissue disorders) | 23 | 12 | 57 | 40
Hand-and-foot syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 7 | 2
Nail disorder (Skin and subcutaneous tissue disorders) | 2 | 1 | 16 | 8
Pruritus (Skin and subcutaneous tissue disorders) | 26 | 15 | 49 | 27
Rash desquamating (Skin and subcutaneous tissue disorders) | 16 | 17 | 42 | 33
Skin disorder (Skin and subcutaneous tissue disorders) | 7 | 3 | 11 | 6
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 | 2 | 7 | 4
Sweating (Skin and subcutaneous tissue disorders) | 5 | 4 | 8 | 1
Hypotension (Vascular disorders) | 10 | 4 | 15 | 10
Thrombosis (Vascular disorders) | 4 | 5 | 7 | 7

LIMITATIONS AND CAVEATS:
Cetuximab arms were added after the study opened, therefore the first 34 patients were excluded from cetuximab analysis. High dose RT arms closed early (at n=474), therefore later patients enrolled to low dose RT arm were excluded from RT analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI's are required to abide by the sponsor's publication guidelines which require review by coauthors and subsequent review and approval by the sponsor.